CLINICAL TRIAL: NCT00857155
Title: Time Based Strategy to Reduce Clopidogrel Associated Bleeding Related to Coronary Artery Bypass Graft (CABG)
Acronym: TARGET-CABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LifeBridge Health (Other)
Responsible Party: Paul A. Gurbel MD, LifeBridge Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB# 1464
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; CABG; Clopidogrel; Aspirin; Point of Care devices
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin only (No Intervention): Continue aspirin until surgery
- Clopidogrel and Aspirin (Other)
  Interventions: Other: Clopidogrel withdraw prior to CABG

INTERVENTIONS:
Other: Clopidogrel withdraw prior to CABG — Patients on clopidogrel are stratified into time-based platelet function recovery groups as determined by point of care methods and based on these groups clopidogrel is withdrawn at a pre-specified timepoint before surgery.
  Arms: Clopidogrel and Aspirin

SUMMARY:
Purpose: In patients with coronary artery disease, aspirin and Plavix are used increasingly to prevent the formation of blood clots in the coronary arteries. These drugs exert their beneficial effects by irreversibly blocking platelets, the compounds found in blood responsible for clotting after an injury or during a heart attack. However, these effects also place patients at increased risk for bleeding after coronary artery bypass surgery. Therefore, it is currently recommended to withhold Plavix therapy for 5 days before undergoing surgery in order to reduce the incidence of bleeding. However, it has been repeatedly shown that Plavix exerts variable effects on different patients, which may be partially explained by poor absorption, drug-drug interaction, and by variations in deoxyribonucleic acid (DNA) which constitutes your genes. In addition, the time required for platelets to regain function after Plavix treatment has been shown to vary between patients. Therefore, by measuring platelet function, it may be possible to determine the optimal amount of time required to withhold Plavix before undergoing bypass surgery, which may improve rates of bleeding following the procedure. The purpose of this study is to classify patients into groups based on platelet function in order to define the ideal time period for delaying surgery. By analyzing the amount of time required for platelet recovery, it is expected that surgery-related bleeding will decrease without increasing the risk of blood clot formation.

Eligibility: Approximately 200 patients requiring CABG will be enrolled at Sinai Hospital, which is the only site where this study is being conducted.

To be eligible you must:

* Be able to provide written informed consent.
* Be between the ages of 18-85 and require CABG.
* Currently be on aspirin therapy (81-325mg).

DETAILED DESCRIPTION:
Primary objective:

We hypothesize that stratifying patients on clopidogrel into time-based platelet function recovery groups as determined by pre-operative clopidogrel response measured by point of care methods will result in similar rates of bleeding as compared to those of clopidogrel naïve patients undergoing elective CABG.

Study design:

This will be a single center, prospective study analyzing clopidogrel naïve patients and patients on clopidogrel with background aspirin therapy requiring CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent.
* Patients must currently be on aspirin therapy (81-325 mg).
* Male or female patients between the ages of 18-85 requiring CABG.

Exclusion Criteria:

* Patients undergoing emergent surgery following failed percutaneous coronary revascularization.
* Patients with a history of previous cardiac surgery and patients needing concomitant valvular surgery.
* Pre-operative exposure to either coumadin or platelet GPIIb/IIIa inhibitors.
* Patients with a history of bleeding diathesis.
* Patients with an activated partial thrombin time >1.5 normal.
* Patients with platelet count <120,000/mm3.
* Patients with hematocrit <30%.
* Patients with creatinine clearance <30mL/min.
* Patients with known active hepatic disease.
* Patients with any other condition that, in the opinion of the investigator, may either put the patient at risk or influence the result of the study (e.g. malignancy, limiting life expectancy, noncompliance).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is chest tube drainage. | During the index hospitalization

SECONDARY OUTCOMES:
The secondary endpoint is transfusion requirements. | Index hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Mahla E, Suarez TA, Bliden KP, Rehak P, Metzler H, Sequeira AJ, Cho P, Sell J, Fan J, Antonino MJ, Tantry US, Gurbel PA. Platelet function measurement-based strategy to reduce bleeding and waiting time in clopidogrel-treated patients undergoing coronary artery bypass graft surgery: the timing based on platelet function strategy to reduce clopidogrel-associated bleeding related to CABG (TARGET-CABG) study. Circ Cardiovasc Interv. 2012 Apr;5(2):261-9. doi: 10.1161/CIRCINTERVENTIONS.111.967208. Epub 2012 Mar 6. PMID 22396581